CLINICAL TRIAL: NCT05676242
Title: A Phase III Extended Clinical Trial of Long-term Safety and Efficacy of Jaktinib Hydrochloride Tablets in the Treatment of Moderate and Severe Atopic Dermatitis
Brief Title: A Phase III Extended Clinical Trial of Jaktinib Hydrochloride Tablets in the Treatment of Moderate and Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK026
Record Dates: First submitted 2022-12-30; First posted 2023-01-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib 100mg BID (Experimental): Drug: Jaktinib Hydrochloride Tablet 100mg dosage, orally administered, twice a day
  Interventions: Drug: Jaktinib Hydrochloride Tablet
- Jaktinib 75mg BID (Experimental): Drug: Jaktinib Hydrochloride Tablet 75mg dosage, orally administered, twice a day
  Interventions: Drug: Jaktinib Hydrochloride Tablet
- Placebo (Placebo Comparator): Drug: Placebo Orally administered, twice a day
  Interventions: Drug: Jaktinib Hydrochloride Tablet

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablet — Orally administered, twice a day

SUMMARY:
To observe the safety and effectiveness of long-term use of jaktinib hydrochloride tablets in the treatment of moderate and severe atopic dermatitis

DETAILED DESCRIPTION:
If the enrolled subjects received the treatment of jaktinib hydrochloride tablets in the ZGJAK025 trial, they will continue to use the drug at the original dosage; If the enrolled subjects received placebo treatment in the ZGJAK025 trial, they will receive 100mg BID of jaktinib hydrochloride tablets, 75mg BID of jaktinib hydrochloride tablets or placebo at a ratio of 1:1:1 at random, and continue to take the drug on an empty stomach, with the longest continuous treatment not exceeding 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The investigator thinks that the subject can continue to benefit from participating in the extension trial;
* Fully understand the extension trial and sign the informed consent form;
* Complete the ZGJAK025 trial for 16 weeks and have good compliance;
* It is expected that the time interval between the first administration and the last administration of ZGJAK025 trial for the subject should be ≤ 4 weeks;

Exclusion Criteria:

* Within 4 weeks before enrollment, there were any adverse events ≥ 3 levels related to the test drug that did not return to level 1 or normal;
* The investigator thinks that the subject is not suitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of subjects with treatment emergent adverse event (TEAE) | 36 weeks after the first dose
  Safety of the drug
Number and percentage of subjects with Serious Adverse Event (SAE) | 36 weeks after the first dose
  Safety of the drug

SECONDARY OUTCOMES:
The diachronic change in the proportion of subjects whose total Eczema area and severity index （EASI） score decreased by ≥ 75% from baseline | 36 weeks after the first dose
  The proportion of subjects who reached EASI-75
The diachronic change of the proportion of subjects whose systemic Investigator's Global Assessment （IGA） score reached 0 or 1 and decreased by ≥ 2 points from baseline | 36 weeks after the first dose
  The proportion of subjects who reached IGA 0/1
The diachronic change in the proportion of subjects whose pruritus Numerical Rating Scale （NRS） score improved by ≥ 4 points from baseline | 36 weeks after the first dose
  The proportion of subjects who reached NRS4

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of Medical Sciences, Peking Union Medical College, Nanjin, Jiangsu

IPD SHARING:
Plan to Share IPD: No